CLINICAL TRIAL: NCT00446186
Title: Mk0476 Phase II Dose Finding Study -Allergic Rhinitis-
Brief Title: MK0476 Study in Adult Patients With Allergic Rhinitis (0476-378)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-378; 2007_009
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Rhinitis Allergic
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — montelukast; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0476, montelukast sodium / Duration of Treatment: 2 Weeks
Drug: Comparator: placebo / Duration of Treatment: 2 Weeks

SUMMARY:
The clinical study evaluates the efficacy and safety of MK0476 in adult patients with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with seasonal allergic rhinitis

Exclusion Criteria:

* Patients who have nasal diseases (e.g., nasal polyp, septonasal arcuation, hypertrophic rhinitis), upper respiratory infection, sinusitis, infectious rhinitis, ocular infection and those disease severe enough to interfere with assessment of effectiveness
* Patients who have rhinitis medicamentosa, or nonallergic rhinitis (e.g., vasomotor rhinitis, eosinophilia rhinitis)
* Patient has a disease of the cardiovascular, hepatic, renal, hematologic systems, or other severe disease

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 945 (Actual)
Dates: Start 2004-02; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
The change from baseline in the composite nasal symptoms score (average over the 2-week treatment period) in seasonal allergic rhinitis

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Okubo K, Baba K. A double-blind non-inferiority clinical study of montelukast, a cysteinyl leukotriene receptor 1 antagonist, compared with pranlukast in patients with seasonal allergic rhinitis. Allergol Int. 2008 Dec;57(4):383-90. doi: 10.2332/allergolint.O-08-533. Epub 2008 Nov 1. PMID 18946234
- [Result] Okubo K, Baba K. Therapeutic effect of montelukast, a cysteinyl leukotriene receptor 1 antagonist, on Japanese patients with seasonal allergic rhinitis. Allergol Int. 2008 Sep;57(3):247-55. doi: 10.2332/allergolint.O-07-515. Epub 2008 Jul 1. PMID 18566548